CLINICAL TRIAL: NCT06154226
Title: Prevention of Post-Cardiac Surgery Acute Kidney Injury by Proton Pump Inhibitor: A Prospective Randomized Controlled Trial
Brief Title: Prevention of Post-Cardiac Surgery Acute Kidney Injury by Proton Pump Inhibitor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Society of Cardiovascular Anesthesiologists (Unknown)
Responsible Party: Principal Investigator, yafen liang, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSC-MS-22-0502
Record Dates: First submitted 2023-11-20; First posted 2023-12-04 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Acute Kidney Injury
Keywords: cardiac surgery
MeSH Terms: conditions — Acute Kidney Injury | interventions — Pantoprazole; Famotidine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor who tests the urinary kidney injury biomarker is blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pantoprazole group (Experimental): Pantoprazole (40 mg iv every 12 hours/q12H) for 2 days perioperatively (first dose after anesthesia induction and before surgical incision, second dose at chest closure, then followed by 2 doses daily (Q12hr dosing) on postoperative (POD) 1 for a total of 4 doses over 2 days. There will be no other modifications in patient care.
  Interventions: Drug: Pantoprazole
- Famotidine Group (Active Comparator): Famotidine (20 mg iv q12H) for 2 days perioperatively (first dose after anesthesia induction and before surgical incision, second dose at chest closure, then followed by 2 doses daily (Q12hr dosing) on POD 1 for a total of 4 doses over 2 days. There will be no other modifications in patient care.
  Interventions: Drug: Famotidine

INTERVENTIONS:
Drug: Pantoprazole — Subjects will receive pantoprazole (40 mg iv q12H) for 2 days perioperatively (first dose after anesthesia induction and before surgical incision, second dose at chest closure, then followed by 2 doses daily (Q12hr dosing) on post operative day 1 (POD 1) for a total of 4 doses over 2 days.
  Arms: Pantoprazole group
Drug: Famotidine — Subjects will receive famotidine (20 mg iv q12H) for 2 days perioperatively (first dose after anesthesia induction and before surgical incision, second dose at chest closure, then followed by 2 doses daily (Q12hr dosing) on POD 1 for a total of 4 doses over 2 days.
  Arms: Famotidine Group

SUMMARY:
The purpose of this study is to determine whether perioperative intravenous administration of pantoprazole will improve kidney function parameters following cardiac surgery with cardiopulmonary bypass compared to famotidine and to determine whether perioperative intravenous administration of pantoprazole will decrease the incidence of postoperative Acte Kidney Injury (AKI) and major adverse kidney events (MAKE).

DETAILED DESCRIPTION:
Each year more than 500,000 cardiac surgeries are performed in the United States of America (USA) alone. Acute kidney injury ( AK) I is a common complication following cardiac surgery and is associated with poor patient outcomes and increased healthcare costs. Therefore, there is an urgent need to identify medical interventions and treatments that prevent AKI or mitigate its severity when it occurs after cardiac surgery.

One of the main causes of AKI following cardiac surgery involves renal hypoperfusion/ischemia and reperfusion injury. Hypoxia-inducible factors (HIFs) are key transcription factors responsible for tissue adaptation to low oxygen, which orchestrate the expression of a wide variety of genes including a set of micro-ribonucleic acid (microRNAs). MicroRNAs are endogenous single-stranded noncoding miRNAs of nucleotides that participate in physiological and pathological functions via regulating post-transcription of target genes. During ischemic injury, hypoxia upregulates endothelial MicroRNAs that has the potential in renal protection through vascular integrity and regeneration. Additionally, microRNAs exert protective effects via decreasing apoptosis and promoting tubular cell proliferation during ischemic AKI.

Moreover, decreased serum levels of MicroRNAs are highly correlated with AKI severity in the intensive care unit (ICU) patients. Our preliminary study identified ATP4A as the downstream target gene of MicroRNAs in the kidney. Adenosine triphosphate (ATP)4A (catalytic α subunit of H+/K+ ATPase) is located in intercalated cells in the distal tubules and cortical collecting ducts, which regulates urine acidification through secretion of hydrogen and reabsorption of potassium from urine. Proton pump inhibitors (PPIs) block the ATP hydrolysis of the H+/K+ ATPase via binding its active site of ATP4A and further enhance this endogenous kidney protection pathway. Despite robust animal model data, randomized controlled trial aiming to test the effectiveness of PPI in post-cardiac surgery AKI prevention is lacking. If proven to be effective, our studies could be easily implemented in clinical practice and serve as an effective treatment for perioperative AKI.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective cardiac surgery with cardio pulmonary bypass (CPB) with a moderate to high risk of developing AKI (Cleveland risk score equal or higher than 3)

Exclusion Criteria:

* Preoperative eGFR<30 ml/min per 1.73 m2
* Dialysis dependence
* Emergency surgery
* Interstitial nephritis
* Pregnancy
* Nursing Patients
* Proton pump inhibitors (PPIs) hypersensitivity
* Liver disease
* Vitamin B12 deficiency

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-09-17 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Kidney Injury Molecule (KIM-1) biomarker changes | Baseline, 8, 24 and 48 hours postoperatively
  Postoperative urinary kidney injury biomarker KIM-1 changes, assessed by the KIM-1 levels at 8, 24, and 48 hours postoperatively adjusted by baseline KIM-1 levels, the speed of KIM-1 changes postoperatively, and the area under the curve (AUC) of KIM-1 levels 24 hours postoperatively

SECONDARY OUTCOMES:
Neutrophil gelatinase-associated lipocalin (NGAL) biomarker changes | Baseline, 8, 24 and 48 hours postoperatively
  Postoperative urinary kidney injury biomarker NGAL changes, assessed by the NGAL levels at 8, 24, and 48 hours postoperatively adjusted by baseline NGAL levels, the speed of NGAL changes postoperatively, and the area under the curve (AUC) of NGAL levels 24 hours postoperatively
Incidence, severity and duration of any-stage postoperative AKI | Post Operative Day 7 (or hospital discharge if earlier).
  AKI will be defined using the 2012 Kidney Disease Improving Global Outcomes (KDIGO) criteria: serum creatinine (SCr) increase greater than 50% from baseline or ≥ 0.3 mg/dL increase within 48 hours after surgery.
Incidence of major adverse kidney events (MAKE) | 30 days after surgery
  MAKE is defined as the composite of death, dialysis, renal hospitalization or sustained kidney dysfunction (glomerular filtration rate/GFR decline of 25% or more from preoperative baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Yafen Liang, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No